CLINICAL TRIAL: NCT07061990
Title: The Role of OSAHS-related Inflammatory Markers in the Pathogenesis of White Matter Lesions and Asymptomatic Lacunar Infarction
Brief Title: The Role of Inflammatory Markers in OSAHS-Related White Matter Lesions and Asymptomatic Lacunar Infarction
Status: Completed | Type: Observational
Sponsor: Yanpeng Li (Other)
Responsible Party: Sponsor-Investigator, Yanpeng Li, Principal investigator, The First Affiliated Hospital of Hebei North University
Organization: The First Affiliated Hospital of Hebei North University (Other)
Other Study IDs: 2022A-34
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Obstructive Sleep Apnea-hypopnea Syndrome
Keywords: OSAHS; Inflammatory Markers; White Matter Lesions; Asymptomatic Lacunar Infarction; Serum Amyloid A (SAA)
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Polysomnography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Simple OSAHS Group: Patients diagnosed with OSAHS who were initially untreated and without a diagnosis of asymptomatic lacunar infarction.
  Interventions: Diagnostic Test: Polysomnography (PSG); Diagnostic Test: Brain Magnetic Resonance Imaging (MRI); Diagnostic Test: Serum Inflammatory Marker Measurement
- Combined Group: Patients diagnosed with OSAHS complicated with asymptomatic lacunar infarction.
  Interventions: Diagnostic Test: Polysomnography (PSG); Diagnostic Test: Brain Magnetic Resonance Imaging (MRI); Diagnostic Test: Serum Inflammatory Marker Measurement
- Control Group: Non-OSAHS individuals who underwent health examinations during the same period and did not have asymptomatic lacunar infarction.
  Interventions: Diagnostic Test: Polysomnography (PSG); Diagnostic Test: Brain Magnetic Resonance Imaging (MRI); Diagnostic Test: Serum Inflammatory Marker Measurement

INTERVENTIONS:
Diagnostic Test: Polysomnography (PSG) — Participants underwent overnight polysomnography for a minimum of 7 hours using an E series polysomnography monitor. The monitoring included electroencephalogram (EEG), eye movement, Holter monitoring, airflow, chest and abdominal respiratory movements, and fingertip oxygen saturation. The results were used to diagnose Obstructive Sleep Apnea-Hypopnea Syndrome (OSAHS) and calculate the Apnea-Hypopnea Index (AHI) for severity classification.
Diagnostic Test: Brain Magnetic Resonance Imaging (MRI) — A whole-brain scan was performed on all participants using a Philips Ingenia 3.0T MRI scanner. The scanning sequences included T1-weighted imaging (T1WI), T2-weighted imaging (T2WI), and Fluid-Attenuated Inversion Recovery (FLAIR). The images were analyzed by two neurologists to identify asymptomatic lacunar infarction and to assess the severity of white matter lesions using the Age-Related White Matter Change (ARWMC) scoring system.
Diagnostic Test: Serum Inflammatory Marker Measurement — Fasting venous blood (3mL) was collected from all participants on the day of their brain MRI scan. Serum was separated by centrifugation. Levels of Serum Amyloid A (SAA), Tumor Necrosis Factor-alpha (TNF-α), and Interleukin-6 (IL-6) were measured using the Enzyme-Linked Immunosorbent Assay (ELISA) method according to the manufacturer's protocols.

SUMMARY:
This retrospective observational study aims to investigate the potential role of inflammatory markers associated with Obstructive Sleep Apnoea-Hypopnoea Syndrome (OSAHS) in the pathogenesis of white matter lesions (WML) and asymptomatic lacunar infarction (ALI). The study compares inflammatory marker levels (SAA, TNF-α, IL-6) and the severity of white matter lesions among patients with OSAHS alone, OSAHS with ALI, and a healthy control group to explore the relationship between the severity of OSAHS, inflammation, and cerebrovascular changes.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea-Hypopnea Syndrome (OSAHS) is a prevalent condition characterized by recurrent upper airway obstruction during sleep, leading to chronic intermittent hypoxia, systemic inflammation, and endothelial dysfunction. These pathological changes are known risk factors for cerebrovascular diseases. White matter lesions and asymptomatic lacunar infarction are early indicators of cerebral small vessel disease and are associated with an increased risk of stroke and cognitive decline. While a link between OSAHS and these brain changes has been suggested, the role of specific inflammatory mediators is not fully understood. This study retrospectively analyzed data from 119 individuals who visited the sleep breathing monitoring clinic between May 2022 and May 2023. Participants were divided into three groups: a simple OSAHS group (n=60), an OSAHS group with concomitant asymptomatic lacunar infarction (combined group, n=29), and a non-OSAHS control group (n=30). The severity of OSAHS was categorized as mild, moderate, or severe based on the Apnea-Hypopnea Index (AHI). The study measured serum levels of Serum Amyloid A (SAA), Tumor Necrosis Factor-alpha (TNF-α), and Interleukin-6 (IL-6). The severity of white matter lesions was assessed using brain MRI and the Age-Related White Matter Change (ARWMC) scoring system. The primary hypothesis is that elevated levels of these OSAHS-related inflammatory markers are associated with the presence and severity of both white matter lesions and asymptomatic lacunar infarction.

ELIGIBILITY:
Inclusion Criteria (for OSAHS and Combined Groups):

* Compliance with the diagnostic criteria for OSAHS (AHI > 5 times/h).
* For Combined Group: Brain MRI or CT evidence of lacunar infarction (diameter ≥3 mm) without a history of acute stroke or neurological deficits.
* No prior OSAHS-related surgery or CPAP treatment.
* Availability of complete clinical data.
* Age > 18 years old.

Inclusion Criteria (for Control Group):

* Did not meet the diagnostic criteria for OSAHS (AHI < 5 times/h).
* No evidence of asymptomatic or symptomatic cerebral infarction.
* Age > 18 years old.

Exclusion Criteria (for all groups):

* Symptomatic cerebral infarction, cerebral hemorrhage, brain injury, or brain tumors.
* Severe anxiety, depression, or other mental illness.
* Severe liver, kidney, heart, or lung dysfunction.
* Acute or chronic infections.
* Other severe respiratory diseases (e.g., COPD, interstitial lung disease).
* Central sleep apnea.
* Coexisting tumor or immune disorders.
* Claustrophobia.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population was sourced from individuals who visited The First Affiliated Hospital of Hebei North University between May 2022 and May 2023. Case participants (patients with OSAHS) were enrolled from the sleep breathing monitoring clinic of the Otolaryngology Department. Control participants were non-OSAHS individuals who underwent health examinations at the same hospital during the same period. All participants were over 18 years old and met detailed inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Levels of Serum Inflammatory Markers | Measured once at the time of enrollment (on the day of brain MRI scan) during the study period from May 2022 to May 2023
  Comparison of serum levels of SAA, TNF-α, and IL-6 among the simple OSAHS group, combined group, and control group.
Correlation between Inflammatory Markers and OSAHS Severity | Measured once at the time of enrollment during the study period from May 2022 to May 2023
  Comparison of SAA, TNF-α, and IL-6 levels across mild, moderate, and severe OSAHS subgroups.
Correlation between Inflammatory Markers and White Matter Lesion Severity | Measured once at the time of enrollment during the study period from May 2022 to May 2023
  Comparison of SAA, TNF-α, and IL-6 levels among patients with normal, mild, and moderate white matter lesions based on ARWMC scores.

SECONDARY OUTCOMES:
Severity of White Matter Lesions | Assessed once via brain MRI at the time of enrollment during the study period from May 2022 to May 2023
  Comparison of the distribution of white matter lesion severity (normal, mild, moderate) among the simple OSAHS group, combined group, and control group.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Hebei North University, Zhangjiakou, Hebei, China